Date: 07/08/2020

**Protocol Version Number: 10** 

Principal Investigator: Jaume Padilla, PhD

**Project IRB #:** 2008181

**Application Title:** Restoring vasodilator actions of insulin in patients with type 2 diabetes (Role of physical activity in restoring vascular insulin sensitivity in skeletal muscle of patients with type 2

diabetes).

**Collaborating Investigators:** 

Elizabeth Parks, PhD Camila Manrique, MD

## **Statistical Analysis Plan**

All statistical analyses were completed with SPSS Statistics (version 23) or GraphPad Prism software (version 8.1.1 or 9.3.0). Statistical comparisons were performed by two-tailed t test or analysis of variance (ANOVA), as appropriate, followed by Tukey's or Bonferroni adjusted pairwise comparisons when significant interactions were found. For all statistical tests, significance was accepted at P<0.05.